CLINICAL TRIAL: NCT07391358
Title: Dual Antiplatelet Therapy Strategy in High Bleeding Risk Patients Undergoing Complex Percutaneous Coronary Intervention Following Acute Coronary Syndrome: Second-Phase Beta Testing of a Patients Decision Aid
Brief Title: DAPT Strategy in HBR Patients Undergoing Complex PCI Following ACS: Second-Phase Beta Testing of a Patients Decision Aid
Acronym: BETA-DAPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Julien Quang Le Van, Pharmacist, Montreal Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2026-3682
Record Dates: First submitted 2026-01-08; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Acute Coronary Syndrome
Keywords: High bleeding risk; Complex percutaneous coronary intervention; Double antiplatelet therapy; Patient decision aid
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High bleeding risk patients treated with complex PCI in the context of ACS (Other): The intervention is the use of the Patient Decision Aid (PDA) to support shared decision-making between patients and clinicians after PCI, assessed using questionnaires capturing multiple dimensions of decision quality.
  No pharmacologic treatment is administered as part of the study; exposure consists solely of complete use of the PDA according to the protocol.
  The study includes a single pre-post group, no interim analyses are planned given the limited project duration, and a single beta-testing phase will be conducted.
  Interventions: Other: Patient decision aid to support shared decision-making between patients and clinicians

INTERVENTIONS:
Other: Patient decision aid to support shared decision-making between patients and clinicians — Patient decision aid to support shared decision-making between patients and clinicians by helping patients understand their risks, available options, and potential consequences, so they can express their preferences regarding antiplatelet therapy.

SUMMARY:
Among patients with acute coronary syndrome (ACS) treated with percutaneous coronary intervention (PCI) and stent implantation, 17.5% are both at high bleeding risk (HBR) and have undergone complex PCI, which also places them at high thrombotic risk. In this population, several dual antiplatelet therapy (DAPT) strategies may be considered: (1) de-escalation of DAPT intensity after 1 to 3 months (switch from ticagrelor/prasugrel to clopidogrel), (2) shortening DAPT duration to 1 to 3 months followed by antiplatelet monotherapy, (3) 12-month clopidogrel-based DAPT, and (4) 12-month ticagrelor/prasugrel-based DAPT. Selecting the most appropriate DAPT strategy in this dual-risk context is complex, and clinical trial evidence is limited for this specific subgroup. In the absence of clear guideline recommendations to support decision-making for patients facing both elevated bleeding and thrombotic risks, structured shared decision-making support is needed.

In this context, within research project 2025-3499 conducted with pharmacy residents, we developed a patient decision aid (PDA) designed to support shared decision-making by helping patients understand their risks, available options, and potential consequences, so they can express their preferences regarding antiplatelet therapy. The PDA aims to facilitate shared decisions by improving patients' understanding of benefits and harms and aligning choices with patient values. A preliminary version of the tool has already undergone alpha testing with a small group of internal users (physicians, pharmacists, and patient partners). The next step is beta testing, that is, real-world testing with the target population and clinicians to evaluate usability and acceptability in routine practice.

ELIGIBILITY:
Inclusion Criteria (Patients)

* Adults aged 18 years or older
* Hospitalized on the coronary care unit ward at the Montreal Heart Institute (MHI)
* Acute coronary syndrome (ACS) during the current episode of care, treated with PCI and placement of one or more coronary stents
* High bleeding risk based on PRECISE-HBR score and high thrombotic risk, with both risks considered of comparable clinical importance by the treating medical team

Inclusion Criteria (Clinicians)

- Clinicians working in the MHI coronary care unit (cardiologists, medical residents, nurse practitioners, or pharmacists) who use the patient decision aid with one or more study participants

Exclusion Criteria (Patients)

* Receiving therapeutic anticoagulation
* Planned cardiac surgery during the same episode of care
* Prior history of coronary stent thrombosis
* Antiphospholipid syndrome or known thrombophilia
* Unable to participate in shared decision-making
* Unable to understand spoken and written French or English
* Concurrent participation in another study (followed within another research protocol)
* Transferred from another center for reasons other than coronary angiography at MHI and expected to return to the referring center for ongoing care (i.e., "fly-in/fly-out" patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Decisional Conflict (DCS-LL) After Use of the Patient Decision Aid (PDA) | Baseline (pre-PDA, Day 0) and immediately post-PDA completion (Day 0, index hospitalization).
  Change in total score on the low-literacy Decisional Conflict Scale (DCS-LL; Ottawa Hospital Research Institute), comparing pre-PDA vs post-PDA completion. Lower scores indicate less decisional conflict.

SECONDARY OUTCOMES:
Change in Antiplatelet Strategy Knowledge Score After PDA Use | Baseline (pre-PDA, Day 0) and immediately post-PDA completion (Day 0, index hospitalization).
  Change in total score on an adapted OHRI knowledge questionnaire assessing understanding of bleeding and thrombotic risks and DAPT options, comparing pre-PDA vs post-PDA completion.
Preparation for Decision-Making (PrepDM) Score After PDA Use | Immediately post-PDA completion (Day 0, index hospitalization).
  Total score on the Preparation for Decision Making (PrepDM; OHRI) questionnaire completed after PDA use. Higher scores indicate greater perceived preparedness to make a decision with the clinician.
Patient Acceptability Score of the PDA in Routine Clinical Use | Immediately post-PDA completion (Day 0, index hospitalization).
  Total score on an OHRI acceptability questionnaire completed after PDA use, reflecting perceived relevance, clarity, length, and overall acceptability in the clinical setting.
Patient Refusal Rate to Use the PDA and Reasons for Refusal | Pre-intervention (at the time of the consent request, prior to PDA delivery, during the index hospitalization).
  Number and proportion of eligible patients who personally refuse participation/PDA use, and categorization of documented reasons for refusal (e.g., not interested, too tired, overwhelmed, language barriers, time constraints).
Agreement Between Patient-Preferred Antiplatelet Strategy and Strategy Prescribed at Hospital Discharge | At hospital discharge (index hospitalization), comparing the patient preference recorded immediately after PDA completion with the antiplatelet strategy on the discharge prescription/orders (also post-PDA completion).
  Proportion of agreement between (a) the antiplatelet strategy preferred by the patient as identified through the PDA and (b) the antiplatelet strategy documented on the discharge prescription/orders.
Clinician Usability of the PDA (French System Usability Scale, F-SUS) | Day 0 (immediately after PDA use with an included patient)
  Total score on the French System Usability Scale (F-SUS) completed by clinicians after using the PDA with an included patient in routine clinical care. Higher scores indicate better usability.
Clinician Refusal Rate to Use the PDA and Reasons for Non-Use | Pre-intervention (at the time the clinician is asked whether it is appropriate to approach the patient and offer the PDA, prior to patient approach and prior to PDA delivery, during the index hospitalization).
  Number and proportion of eligible patient encounters in which the clinician declines to use the PDA when asked, along with categorization of documented reasons (e.g., time constraints, clinical instability, workflow barriers, clinician preference).

OTHER OUTCOMES:
Exploratory Subgroup Effects on Decisional Conflict Scores Low Litteracy (DCS-LL) Questionnaire | Baseline (pre-PDA, Day 0) and immediately post-PDA completion (Day 0, index hospitalization).
  Exploratory assessment of whether changes in DCS-LL differ by prespecified characteristics: age (<70 vs ≥70 years), sex (male vs female), mother tongue (French vs English), education level (university vs lower) and prior percutaneous intervention with stent (yes or no). Analyses are descriptive/exploratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No